CLINICAL TRIAL: NCT02696382
Title: Improving Function in Older Veterans With Hospital-associated Deconditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E1978-R; 15-1571 (Other: VA Eastern Colorado Health Care System)
Record Dates: First submitted 2016-02-19; First posted 2016-03-02 (Estimated); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-09

CONDITIONS: Frail Elderly; Homebound Persons
Keywords: Veterans; Progressive High Intensity Physical Therapy; Gait Speed; Acute Hospitalization; Hospital Associated Deconditioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (UC) (Active Comparator): Participants in the "Usual Care" (UC) group will receive standard, low-intensity physical therapy following discharge from acute hospitalization.
  Interventions: Behavioral: Usual Care (UC)
- Progressive High Intensity Therapy (Experimental): Participants in the "Progressive High Intensity Therapy" (PHIT) group will receive high intensity physical therapy following discharge from acute hospitalization.
  Interventions: Behavioral: Progressive High Intensity Therapy (PHIT)

INTERVENTIONS:
Behavioral: Progressive High Intensity Therapy (PHIT) — Participants in the "Progressive High Intensity Therapy" (PHIT) group will receive high intensity physical therapy following discharge from acute hospitalization. The activities of training will include progressive resistance training, multi-planar motor control and gait exercises, and high intensity activities of daily living training. Like the Usual Care group, the PHIT participants will receive 12 intervention visits over 4 weeks (3 visits per week). Participants will also receive a standardized home exercise program.
  Arms: Progressive High Intensity Therapy
Behavioral: Usual Care (UC) — Participants in the "Usual Care" group will receive standard physical therapy following discharge from acute hospitalization. The activities of therapy will include basic strength training, single-planar motor control and gait exercises, and activities of daily living training. Participants will receive 12 intervention visits over 4 weeks (3 visits per week). Participants will also receive a standardized home exercise program.
  Arms: Usual Care (UC)

SUMMARY:
The investigators plan to test an innovative, home-based, short duration, high intensity exercise program designed for application in the immediate post-hospitalization period in older Veterans. Preliminary data suggest a more intensive approach to physical therapy in older adults after hospitalization is safe and maximizes mobility more than usual care. The Veterans participating in the high intensity exercise program will receive therapy utilizing higher resistance exercises. Outcomes from this group will be compared to data collected from the patients receiving standard, lower resistance therapies.

DETAILED DESCRIPTION:
Hospital associated deconditioning is a common and profound contributor to functional decline in older adults. Skeletal muscle weakness and atrophy are commonly observed in older adults with deconditioning after a hospitalizations, leading to chronic functional deficits. This is especially concerning for elderly Veterans, a population who tends to suffer from more chronic conditions and have decreased physical function than the general older adult population. Therefore, Veterans may be at even higher risk for developing disability in activities of daily living after hospitalization and be homebound. Home health physical therapy may be the ideal venue for addressing this functional decline as around 3 million older adults receive home health services following hospital discharge. These services, however, tend to be low intensity and do not appear to adequately address deficits in function or performance of home and community mobility. To address these concerns, the investigators have developed and tested an innovative, short-duration, home-based, high intensity exercise program designed for application immediately following hospitalization. This protocol will dose twelve therapy visits over the course of 30 days to determine whether visit frontloading has any effect on outcomes. The investigators are using a series of high resistance therapy exercises following acute hospitalization to determine if progressive high intensity therapy sustainability improves physical function more than standard home health physical therapy after an acute hospitalization in older Veterans. Outcomes will spotlight physical function, community mobility, Activities of Daily Living, quality of life, and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Recent hospitalization or period of deconditioning
* Veteran Status
* Referred to or eligible for home health physical therapy
* Have at least 3 comorbid conditions including: Chronic Obstructive Pulmonary Disease (COPD), pneumonia, hypertension, hernia, heart disease, spinal stenosis, atrial fibrillation, post-op bowel surgery, gastrointestinal bleed, chronic ulcerative wounds, depression/ mental health, post-op pancreatic surgery, hypercholesterolemia, dehydration, hypo/hyperthyroid, congestive heart failure, urinary tract infection, diabetes, irritable bowel syndrome, osteoporosis, osteoarthritis, rheumatoid arthritis, gout, peripheral artery disease, syncope, renal failure-no dialysis
* Be ambulatory without human assistance prior to hospitalization

Exclusion Criteria:

* Acute lower extremity fracture with weight-bearing restriction
* Elective joint replacement surgery
* Lower extremity amputation
* Acute cardiac surgery
* Terminal illness
* Cancer
* Alzheimer's disease
* Deep vein thrombosis
* Recent stroke

  * Degenerative neurological conditions
  * Gait speed slower than 0.3 m/s or >1.0 meters/second
* Inability to walk 10 feet without human assistance --History of illegal substance use

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Stevens-Lapsley, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mangione KK, Lopopolo RB, Neff NP, Craik RL, Palombaro KM. Interventions used by physical therapists in home care for people after hip fracture. Phys Ther. 2008 Feb;88(2):199-210. doi: 10.2522/ptj.20070023. Epub 2007 Dec 4. PMID 18056752
- [Background] Falvey JR, Mangione KK, Stevens-Lapsley JE. Rethinking Hospital-Associated Deconditioning: Proposed Paradigm Shift. Phys Ther. 2015 Sep;95(9):1307-15. doi: 10.2522/ptj.20140511. Epub 2015 Apr 23. PMID 25908526
- [Background] Tinetti ME, Baker D, Gallo WT, Nanda A, Charpentier P, O'Leary J. Evaluation of restorative care vs usual care for older adults receiving an acute episode of home care. JAMA. 2002 Apr 24;287(16):2098-105. doi: 10.1001/jama.287.16.2098. PMID 11966384
- [Background] Andersen LL, Andersen CH, Mortensen OS, Poulsen OM, Bjornlund IB, Zebis MK. Muscle activation and perceived loading during rehabilitation exercises: comparison of dumbbells and elastic resistance. Phys Ther. 2010 Apr;90(4):538-49. doi: 10.2522/ptj.20090167. Epub 2010 Feb 4. PMID 20133444
- [Background] El Solh A, Pineda L, Bouquin P, Mankowski C. Determinants of short and long term functional recovery after hospitalization for community-acquired pneumonia in the elderly: role of inflammatory markers. BMC Geriatr. 2006 Aug 9;6:12. doi: 10.1186/1471-2318-6-12. PMID 16899118

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 90 post-consent screen failures
Groups:
- Usual Care (UC): Participants in the "Usual Care" (UC) group received standard, low-intensity physical therapy following discharge from acute hospitalization.
  Usual Care (UC): Participants in the "Usual Care" group received standard physical therapy following discharge from acute hospitalization. The activities of therapy included basic strength training, single-planar motor control and gait exercises, and activities of daily living training. Participants received 12 intervention visits over 4 weeks (3 visits per week). Participants also received a standardized home exercise program.
- Progressive High Intensity Therapy: Participants in the "Progressive High Intensity Therapy" (PHIT) group received high intensity physical therapy following discharge from acute hospitalization.
  Progressive High Intensity Therapy (PHIT): Participants in the "Progressive High Intensity Therapy" (PHIT) group received high intensity physical therapy following discharge from acute hospitalization. The activities of training included progressive resistance training, multi-planar motor control and gait exercises, and high intensity activities of daily living training. Like the Usual Care group, the PHIT participants received 12 intervention visits over 4 weeks (3 visits per week). Participants also received a standardized home exercise program.
Period: Overall Study
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Started | 75 | 75
30-Day Assessment | 65 | 69
60-Day Assessment | 64 | 66
90-Day Assessment | 63 | 64
Completed | 59 | 54
Not Completed | 16 | 21
Not completed — Death | 7 | 2
Not completed — Withdrawal by Subject | 5 | 12
Not completed — Lost to Follow-up | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Median (Full Range); unit: Years] | 76.0 [56 to 95] | 77.0 [59 to 93] | 76.5 [56 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 17 | 23
  Male | 69 | 58 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 14 | 21
  Not Hispanic or Latino | 63 | 59 | 122
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 18 | 28
  White | 58 | 50 | 108
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75 | 75 | 150
Education [Count of Participants; unit: Participants]
  Less Than High School | 5 | 3 | 8
  High School Diploma | 17 | 23 | 40
  Some College | 21 | 26 | 47
  Associate's | 10 | 8 | 18
  Bachelor's/Master's/Doctoral | 21 | 15 | 36
  Unknown or Not Reported | 1 | 0 | 1
Marital Status [Count of Participants; unit: Participants]
  Single | 6 | 9 | 15
  Married/Cohabitating | 29 | 33 | 62
  Widowed | 13 | 16 | 29
  Divorced/Separated | 18 | 16 | 34
  Unknown or Not Reported | 9 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-Selected Walking Speed
Description: Will be assessed at the subject's self selected speed for each participant over 4 meters. Faster walking indicates capacity for performance of certain activities (e.g. crossing a street before the light changes).
Time Frame: From baseline to 60 days post-baseline
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 58 | 59
m/s | 0.08 [0.04 to 0.12] | 0.08 [0.04 to 0.12]

2. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: The SPPB is a well-accepted global measure of lower extremity function which consists of a composite measure including walking speed, chair stands, and balance. It is a strong predictor of disability, institutionalization, and morbidity in older adults. The SPPB is comprised of 3 tasks: a hierarchical standing balance test (side-by-side, semi-tandem, and tandem), a 4-meter usual gait speed, and a 5-time sit-to-stand from a standardized chair. Each subtask is scored (based on time) from 0-4 points and then summarized into a total score of 0-12 points, where 12 points represents the highest performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 73 | 74
score on a scale | 5.07 (2.50) | 5.27 (2.54)

3. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: as for outcome 2
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 61 | 64
score on a scale | 6.46 (3.13) | 6.22 (2.86)

4. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: as for outcome 2
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 60 | 61
score on a scale | 6.50 (3.30) | 6.11 (3.15)

5. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: as for outcome 2
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 58 | 60
score on a scale | 6.43 (3.27) | 5.97 (3.05)

6. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: as for outcome 2
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 57 | 52
score on a scale | 6.82 (3.30) | 6.46 (3.16)

7. Secondary Outcome: Timed-Up-And-Go Test
Description: The TUG measures the time it takes a patient to rise from an arm chair (seat height of 46 cm), walk 3 m, turn and return to sitting in the same chair without physical assistance. This test has excellent inter-rater (ICC=0.99) and intra-rater reliability (ICC=0.99), as measured in a group of 60 functionally disabled older adults (mean age 80 years). Faster times indicate a better outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 67 | 65
seconds | 22.91 (18.74) | 19.98 (11.81)

8. Secondary Outcome: Timed-Up-And-Go Test
Description: as for outcome 7
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 55 | 60
seconds | 16.15 (9.67) | 16.15 (7.61)

9. Secondary Outcome: Timed-Up-And-Go Test
Description: as for outcome 7
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 53 | 52
seconds | 18.47 (15.32) | 17.21 (9.56)

10. Secondary Outcome: Timed-Up-And-Go Test
Description: as for outcome 7
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 54 | 52
seconds | 18.80 (3.27) | 17.78 (14.14)

11. Secondary Outcome: Timed-Up-And-Go Test
Description: as for outcome 7
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 49 | 45
seconds | 15.96 (8.26) | 16.61 (9.73)

12. Secondary Outcome: Modified Physical Performance Test (mPPT)
Description: mPPT assesses 7 tasks. Based on the time it takes to complete each task, a score from 0 (unable to complete) to 4 (performed quickly and easily) is given for each item. The maximal score is 28 and includes tasks that involve upper and lower extremity function. Test-retest reliability for the modified PPT score is 0.96. The instrument is sensitive to change and has been used in exercise trials with frail elders.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 71 | 72
score on a scale | 12.31 (6.57) | 12.08 (6.29)

13. Secondary Outcome: Modified Physical Performance Test (mPPT)
Description: as for outcome 12
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 58 | 62
score on a scale | 16.47 (7.43) | 15.37 (6.88)

14. Secondary Outcome: Modified Physical Performance Test (mPPT)
Description: as for outcome 12
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 57 | 55
score on a scale | 16.04 (7.60) | 15.38 (6.61)

15. Secondary Outcome: Modified Physical Performance Test (mPPT)
Description: as for outcome 12
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 56 | 56
score on a scale | 15.63 (7.32) | 15.07 (7.4)

16. Secondary Outcome: Modified Physical Performance Test (mPPT)
Description: as for outcome 12
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 55 | 47
score on a scale | 15.49 (7.77) | 16.51 (7.07)

17. Secondary Outcome: Lower Extremity Strength Via Hand-Held Dynamometry: Right Knee Extensor
Description: Quadriceps muscle strength was tested via hand-held dynamometry (Lafayette Instrument Company, Lafayette, IN), wherein higher numbers indicate greater strength (better outcome). Method established in previous work: The position of the dynamometer was held perpendicular to the limb segment toward which it was directed, and the plate of the dynamometer was placed in the same position on the tested limb each time. The tester manually stabilized the limb segment proximally and provided verbal and visual cues of the muscle contraction prior to the isometric test. Individuals were asked to maintain the maximum effort for 2-3 seconds, at which point the tester told them to stop. Strength for each muscle was tested until two maximal attempts were within 5% of each other, and the highest value, to the nearest tenth of a kg, was used in analysis.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 52 | 54
kg | 19.03 (9.32) | 18.08 (9.10)

18. Secondary Outcome: Lower Extremity Strength Via Hand-Held Dynamometry: Right Knee Extensor
Description: as for outcome 17
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 49 | 53
kg | 18.67 (6.12) | 19.09 (10.07)

19. Secondary Outcome: Lower Extremity Strength Via Hand-Held Dynamometry: Right Knee Extensor
Description: as for outcome 17
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 45 | 48
kg | 21.11 (9.04) | 18.61 (6.80)

20. Secondary Outcome: Lower Extremity Strength Via Hand-Held Dynamometry: Right Knee Extensor
Description: as for outcome 17
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 41 | 43
kg | 19.24 (7.57) | 19.34 (5.13)

21. Secondary Outcome: Lower Extremity Strength Via Hand-Held Dynamometry: Right Knee Extensor
Description: as for outcome 17
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 40 | 37
kg | 20.99 (7.76) | 19.37 (7.18)

22. Secondary Outcome: Lower Extremity Strength Via Hand-Held Dynamometry: Left Knee Extensor
Description: as for outcome 17
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 51 | 52
kg | 18.64 (8.23) | 18.73 (10.54)

23. Secondary Outcome: Lower Extremity Strength Via Hand-Held Dynamometry: Left Knee Extensor
Description: as for outcome 17
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 49 | 51
kg | 18.17 (6.28) | 19.80 (10.28)

24. Secondary Outcome: Lower Extremity Strength Via Hand-Held Dynamometry: Left Knee Extensor
Description: as for outcome 17
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 46 | 47
kg | 20.52 (8.29) | 18.13 (7.16)

25. Secondary Outcome: Lower Extremity Strength Via Hand-Held Dynamometry: Left Knee Extensor
Description: as for outcome 17
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 42 | 43
kg | 17.74 (6.72) | 18.93 (6.55)

26. Secondary Outcome: Lower Extremity Strength Via Hand-Held Dynamometry: Left Knee Extensor
Description: as for outcome 17
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 39 | 36
kg | 19.86 (6.57) | 19.52 (7.91)

27. Secondary Outcome: Grip Strength: Dominant Hand
Description: Grip strength was measured on the dominant hand using a hand dynamometer with the participant seated and elbow positioned at 90 degrees of flexion with the arm resting against the trunk. Maximal grip strength during a 3 second hold was measured for at least 2 trials and a 3rd trial was allowed if differences between trials were > 5%. Higher numbers indicate greater strength (better outcome).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 66 | 64
kg | 24.60 (8.98) | 27.94 (13.10)

28. Secondary Outcome: Grip Strength: Dominant Hand
Description: as for outcome 27
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 58 | 62
kg | 26.06 (9.34) | 26.21 (11.31)

29. Secondary Outcome: Grip Strength: Dominant Hand
Description: as for outcome 27
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 58 | 59
kg | 26.57 (8.70) | 25.81 (10.77)

30. Secondary Outcome: Grip Strength: Dominant Hand
Description: as for outcome 27
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 55 | 56
kg | 26.13 (7.22) | 27.35 (11.75)

31. Secondary Outcome: Grip Strength: Dominant Hand
Description: as for outcome 27
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 50 | 51
kg | 26.15 (8.03) | 27.86 (10.98)

32. Secondary Outcome: Self-Selected Walking Speed
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 73 | 74
m/s | 0.49 (0.19) | 0.50 (0.17)

33. Secondary Outcome: Self-Selected Walking Speed
Description: as for outcome 1
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 59 | 65
m/s | 0.59 (0.20) | 0.57 (0.22)

34. Secondary Outcome: Self-Selected Walking Speed
Description: as for outcome 1
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 59 | 59
m/s | 0.61 (0.22) | 0.60 (0.27)

35. Secondary Outcome: Self-Selected Walking Speed
Description: as for outcome 1
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 57 | 52
m/s | 0.63 (0.24) | 0.60 (0.23)

36. Other Pre Specified Outcome: Patient Activation Measure Survey (PAM)
Description: A self-administered, validated survey identifying patient motivation levels regarding their healthcare. The PAM survey can reliably predict ER visits, hospital admissions, and medication/ therapy adherence. The final score is a composite score of the available 13 items, ranging from 0-100, wherein a higher score indicates a higher activation (better outcomes).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 69 | 71
score on a scale | 60.82 (13.04) | 62.13 (14.04)

37. Other Pre Specified Outcome: Step Count
Description: Mounted, tri-axial accelerometer activPAL (PAL Technologies Ltd, Glasgow, UK) was used to capture steps. The activPAL was mounted following completion of the associated assessment and was set to record physical activity for a 24-hour/day, 10-day wear protocol. Data was analyzed with the CREA algorithm (PAL Technologies Ltd) to determine valid wear days. Average step count across valid wear days was used for analysis.
Time Frame: Baseline
Population: Activity monitor placement was deferred for those participants who declined placement, demonstrated impaired skin integrity, or were unable to understand instructions.
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 45 | 53
steps per day | 2298.56 (1774.04) | 2190.65 (1367.09)

38. Other Pre Specified Outcome: Step Count
Description: as for outcome 37
Time Frame: 60 Days
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 34 | 36
steps per day | 3098.33 (2125.86) | 2724.17 (1675.40)

39. Other Pre Specified Outcome: Step Count
Description: as for outcome 37
Time Frame: 180 Days
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 30 | 32
steps per day | 2410.59 (1737.08) | 2583.33 (1403.92)

40. Other Pre Specified Outcome: The Life-Space Assessment Survey
Description: The Life-Space Assessment survey is a self-reported measure assessing a patient's movement, extending from within the home to beyond a patient's town or geographic region during the prior 4 weeks. The composite score (summed) ranges from 0 to 120, with higher scores representing greater mobility.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 62 | 63
score on a scale | 34.01 (16.43) | 32.13 (16.69)

41. Other Pre Specified Outcome: The Life-Space Assessment Survey
Description: as for outcome 40
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 57 | 58
score on a scale | 39.79 (15.75) | 39.71 (15.91)

42. Other Pre Specified Outcome: The Life-Space Assessment Survey
Description: as for outcome 40
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 59 | 56
score on a scale | 40.92 (41.56) | 38.71 (19.99)

43. Other Pre Specified Outcome: The Life-Space Assessment Survey
Description: as for outcome 40
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 53 | 57
score on a scale | 41.57 (16.70) | 40.54 (17.61)

44. Other Pre Specified Outcome: The Life-Space Assessment Survey
Description: as for outcome 40
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 54 | 45
score on a scale | 42.62 (20.40) | 40.17 (39.00)

45. Other Pre Specified Outcome: The Veterans Rand 12 Items Health Survey (VR-12): Physical Component Score (PCS)
Description: The Veterans RAND 12 Item Health Survey (VR-12) is a patient-reported global health measure that is used to assess a patient's overall perspective of their health. The questions in this survey correspond to seven different health domains: general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy/fatigue levels, social functioning and mental health. Answers are summarized into two scores, a Physical Component Score (PCS) and a Mental Component Score (MCS) which then provides an important contrast between the respondents' physical and psychological health status. Each component score is summarized from 0 to 100, with a higher score indicating a better outcome.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 72 | 74
score on a scale | 29.34 (8.64) | 28.82 (9.29)

46. Other Pre Specified Outcome: The Veterans Rand 12 Items Health Survey (VR-12): Physical Component Score (PCS)
Description: as for outcome 45
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 61 | 60
score on a scale | 32.94 (10.28) | 32.41 (11.58)

47. Other Pre Specified Outcome: The Veterans Rand 12 Items Health Survey (VR-12): Physical Component Score (PCS)
Description: as for outcome 45
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 54 | 49
score on a scale | 33.77 (10.80) | 32.55 (10.60)

48. Other Pre Specified Outcome: The Veterans Rand 12 Items Health Survey (VR-12): Mental Component Score (MCS)
Description: as for outcome 45
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 72 | 73
score on a scale | 45.83 (12.34) | 45.03 (12.94)

49. Other Pre Specified Outcome: The Veterans Rand 12 Items Health Survey (VR-12): Mental Component Score (MCS)
Description: as for outcome 45
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 60 | 60
score on a scale | 48.83 (12.91) | 45.30 (15.04)

50. Other Pre Specified Outcome: The Veterans Rand 12 Items Health Survey (VR-12): Mental Component Score (MCS)
Description: as for outcome 45
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 54 | 49
score on a scale | 50.70 (11.53) | 44.13 (12.36)

51. Other Pre Specified Outcome: St. Louis University Mental Status Examination (SLUMS)
Description: SLUMS screens for cognitive impairments by assessing participant function in the areas of attention, calculation, immediate and delayed recall, animal naming, and visuospatial skills. Scores range from 0 to 30, wherein a higher score indicates less cognitive impairment. Scores of 27 to 30 are considered normal in a person with a high school education. Scores between 21 and 26 suggest a mild neurocognitive disorder. Scores between 0 and 20 indicate dementia.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 71 | 74
score on a scale | 22.68 (4.14) | 22.28 (4.30)

52. Other Pre Specified Outcome: St. Louis University Mental Status Examination (SLUMS)
Description: as for outcome 51
Time Frame: 60 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 58 | 59
score on a scale | 23.17 (4.78) | 22.49 (4.78)

53. Other Pre Specified Outcome: St. Louis University Mental Status Examination (SLUMS)
Description: as for outcome 51
Time Frame: 180 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
Number analyzed (Participants) | 51 | 49
score on a scale | 23.86 (4.40) | 22.59 (5.01)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment to 6 months following baseline assessment.
Description: Adverse events were collected via questionnaire every 30 days for 180 days following baseline assessment. The questionnaire included questions regarding expected adverse events: falls, ED visits, and hospitalizations.
Arm/Group | Usual Care (UC) | Progressive High Intensity Therapy
All-Cause Mortality (participants affected / at risk) | 7/75 | 2/75
Serious Adverse Events (participants affected / at risk) | 33/75 | 34/75
Other Adverse Events (participants affected / at risk) | 46/75 | 47/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (UC) (N=75) | Progressive High Intensity Therapy (N=75)
Death (General disorders) | 7 (7) | 2 (2)
Inpatient Hospitalization (General disorders) | 30 (54) | 33 (49)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (UC) (N=75) | Progressive High Intensity Therapy (N=75)
Falls (General disorders) | 35 (82) | 31 (91)
ED Visit Not Requiring Hospitalization (General disorders) | 33 (53) | 30 (58)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT02696382/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT02696382/ICF_001.pdf